CLINICAL TRIAL: NCT04988646
Title: Pharmacokinetic Properties of Acyclovir
Brief Title: Pharmacokinetic Properties of 200 and 400 mg Acyclovir Tablet in Indonesia Healthy Subject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT. Kimia Farma (Persero) Tbk (Industry)
Collaborators: PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 515/STD/PML/2019
Record Dates: First submitted 2021-07-06; First posted 2021-08-03 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Drug Use
Keywords: bioequivalence; pharmacokinetics; Indonesian healthy subject; Acyclovir
MeSH Terms: interventions — Acyclovir; Tablets

STUDY DESIGN:
Intervention Model Description: Randomized, single blind, single dose, 2-periods, cross-over design study with one week washout period between each treatment in 28 healthy subjects under fasting condition
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acyclovir Tablet (Experimental): Participants received Acyclovir Tablet 200 mg or 400 mg with 240 mL of water
  Interventions: Drug: Acyclovir 200 MG; Drug: Acyclovir 400 MG
- Zovirax® Tablet (Active Comparator): Participants received Zovirax® Tablet 200 mg or 2x200 mg with 240 mL of water
  Interventions: Drug: Zovirax 200 MG Tablet; Drug: Zovirax 400 MG Tablet

INTERVENTIONS:
Drug: Acyclovir 200 MG — Administered with 240 mL of water
  Arms: Acyclovir Tablet
Drug: Acyclovir 400 MG — Administered with 240 mL of water
  Arms: Acyclovir Tablet
Drug: Zovirax 200 MG Tablet — Administered with 240 mL of water
  Arms: Zovirax® Tablet
Drug: Zovirax 400 MG Tablet — Administered with 240 mL of water
  Arms: Zovirax® Tablet

SUMMARY:
The objective of this present study was to asses the pharmacokinetic properties of acyclovir tablet from new product formulation (PT. Kimia Farma (Persero) Tbk) to its innovator product, Zovirax® tablet (Glaxo Wellcome S.A., Aranda, Spain)

DETAILED DESCRIPTION:
Twenty-eight healty subjects were given a single dose of acyclovir tablet or Zovirax® in dosage form 200 mg and 400mg with 240 mL of water. Then the blood samples for acyclovir was drawn and analyzed using LCMS/MS. All subjects sample plasma were analyzed for pharmacokinetic evaluation

ELIGIBILITY:
Inclusion Criteria:

* body weight within normal range (body mass index between 18 and 25 kg/m2)
* had normal blood pressure (systolic was ranged between 90 to 120 mmHg and diastolic was ranged between 60 to 80 mmHg)
* had normal electrocardiogram
* absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening

Exclusion Criteria:

* pregnant women
* nursing mothers
* women of childbearing potential without adequate contraception
* had a history of contraindication or hypersensitivity to aciclovir, or other antiviral or other ingredients in the study products or a history of serious allergic reaction to any drug,
* a significant allergic disease, or allergic reaction; presence of medical condition which might significantly influence the pharmacokinetics of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction or cardiovascular disease
* presence of any coagulation disorder or clinically significant hematology abnormalities; using any medication (prescription or non-prescription drug, food supplement, herbal medicine)
* particularly the medication known to affect the pharmacokinetics of the study drug
* who had participated in any clinical study within 3 months prior to the study (< 90 days)
* subjects who had donated or lost 300 ml (or more) of blood within 3 months prior to the study
* who were positive to HIV, HBsAg, and HCV tests
* who were unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits
* poor venous access; and who smoked more than 10 cigarettes a day
* had a history of drug or alcohol abuse within 12 months prior to screening for this study and who were unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits, poor venous access

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Metta Sinta Sari Wiria, Principal Investigator — PT Pharma Metric Labs; I Gusti Putu Bagus Diana Virgo, Study Director — PT Pharma Metric Labs
Locations (1):
- PT Pharma Metric Labs, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Result] Stahl JP, Mailles A. Herpes simplex virus encephalitis update. Curr Opin Infect Dis. 2019 Jun;32(3):239-243. doi: 10.1097/QCO.0000000000000554. PMID 30921087
- [Result] Ahronowitz I, Fox LP. Herpes zoster in hospitalized adults: Practice gaps, new evidence, and remaining questions. J Am Acad Dermatol. 2018 Jan;78(1):223-230.e3. doi: 10.1016/j.jaad.2017.07.054. Epub 2017 Nov 14. PMID 29146146
- [Result] Kukhanova MK, Korovina AN, Kochetkov SN. Human herpes simplex virus: life cycle and development of inhibitors. Biochemistry (Mosc). 2014 Dec;79(13):1635-52. doi: 10.1134/S0006297914130124. PMID 25749169
- [Result] Vaithianathan S, Haidar SH, Zhang X, Jiang W, Avon C, Dowling TC, Shao C, Kane M, Hoag SW, Flasar MH, Ting TY, Polli JE. Effect of Common Excipients on the Oral Drug Absorption of Biopharmaceutics Classification System Class 3 Drugs Cimetidine and Acyclovir. J Pharm Sci. 2016 Feb;105(2):996-1005. doi: 10.1002/jps.24643. Epub 2016 Jan 12. PMID 26375604
- [Result] de Miranda P, Blum MR. Pharmacokinetics of acyclovir after intravenous and oral administration. J Antimicrob Chemother. 1983 Sep;12 Suppl B:29-37. doi: 10.1093/jac/12.suppl_b.29. PMID 6355048
- [Result] O'Brien JJ, Campoli-Richards DM. Acyclovir. An updated review of its antiviral activity, pharmacokinetic properties and therapeutic efficacy. Drugs. 1989 Mar;37(3):233-309. doi: 10.2165/00003495-198937030-00002. PMID 2653790
- [Result] Fletcher C, Bean B. Evaluation of oral acyclovir therapy. Drug Intell Clin Pharm. 1985 Jul-Aug;19(7-8):518-24. doi: 10.1177/106002808501900703. PMID 2992899
- [Result] Al-Yamani MJ, Al-Khamis KI, El-Sayed YM, Bawazir SA, Al-Rashood KA, Gouda MW. Comparative bioavailability of two tablet formulations of acyclovir in healthy volunteers. Int J Clin Pharmacol Ther. 1998 Apr;36(4):222-6. PMID 9587049
- [Result] Amini H, Javan M, Gazerani P, Ghaffari A, Ahmadiani A. Lack of bioequivalence between two aciclovir tablets in healthy subjects. Clin Drug Investig. 2008;28(1):47-53. doi: 10.2165/00044011-200828010-00006. PMID 18081360
- [Result] Weller S, Blum MR, Doucette M, Burnette T, Cederberg DM, de Miranda P, Smiley ML. Pharmacokinetics of the acyclovir pro-drug valaciclovir after escalating single- and multiple-dose administration to normal volunteers. Clin Pharmacol Ther. 1993 Dec;54(6):595-605. doi: 10.1038/clpt.1993.196. PMID 8275615
- [Result] Galgatte UC, Jamdade VR, Aute PP, Chaudhari PD. Study on requirements of bioequivalence for registration of pharmaceutical products in USA, Europe and Canada. Saudi Pharm J. 2014 Nov;22(5):391-402. doi: 10.1016/j.jsps.2013.05.001. Epub 2013 May 31. PMID 25473327
- [Result] Corrao G, Soranna D, La Vecchia C, Catapano A, Agabiti-Rosei E, Gensini G, Merlino L, Mancia G. Medication persistence and the use of generic and brand-name blood pressure-lowering agents. J Hypertens. 2014 May;32(5):1146-53; discussion 1153. doi: 10.1097/HJH.0000000000000130. PMID 24569417
- [Result] Kesselheim AS, Misono AS, Lee JL, Stedman MR, Brookhart MA, Choudhry NK, Shrank WH. Clinical equivalence of generic and brand-name drugs used in cardiovascular disease: a systematic review and meta-analysis. JAMA. 2008 Dec 3;300(21):2514-26. doi: 10.1001/jama.2008.758. PMID 19050195

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted with two types of drug doses, which were dose of 200 mg and 400 mg. Of each dose performed on 28 subjects
Groups:
- Test Drug First, Then Reference Drug for Dose 200 mg: Participants received New (test) Acyclovir Tablet 200 mg with 240 mL of water as a single oral dose in the first intervention period, and marketed (reference) Zovirax® 200 mg Tablet with 240 mL of water as a single oral dose in the second intervention period (after washout period).
- Reference Drug First, Then Test Drug for Dose 200 mg: Participants received marketed (reference) Zovirax® 200 mg Tablet with 240 mL of water as a single oral dose in the first intervention period, and new (test) Acyclovir 200 mg Tablet with 240 mL of water as a single oral dose in the second intervention period (after washout period).
- Test Drug First, Then Reference Drug for Dose 400 mg: Participants received New (test) Acyclovir Tablet 400 mg with 240 mL of water as a single oral dose in the first intervention period, and marketed (reference) Zovirax® 2x200 mg Tablet with 240 mL of water as a single oral dose in the second intervention period (after washout period).
- Reference Drug First, Then Test Drug for Dose 400 mg: Participants received marketed (reference) Zovirax® 2x200 mg Tablet with 240 mL of water as a single oral dose in the first intervention period, and new (test) Acyclovir 400 mg Tablet with 240 mL of water as a single oral dose in the second intervention period (after washout period).
Period: 1st Intervention
Arm/Group | Test Drug First, Then Reference Drug for Dose 200 mg | Reference Drug First, Then Test Drug for Dose 200 mg | Test Drug First, Then Reference Drug for Dose 400 mg | Reference Drug First, Then Test Drug for Dose 400 mg
Started | 14 | 14 | 14 | 14
Completed | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Washout >= One Week
Arm/Group | Test Drug First, Then Reference Drug for Dose 200 mg | Reference Drug First, Then Test Drug for Dose 200 mg | Test Drug First, Then Reference Drug for Dose 400 mg | Reference Drug First, Then Test Drug for Dose 400 mg
Started | 14 | 14 | 14 | 14
Completed | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0
Period: 2nd Intervention
Arm/Group | Test Drug First, Then Reference Drug for Dose 200 mg | Reference Drug First, Then Test Drug for Dose 200 mg | Test Drug First, Then Reference Drug for Dose 400 mg | Reference Drug First, Then Test Drug for Dose 400 mg
Started | 14 | 14 | 14 | 14
Completed | 13 | 13 | 14 | 14
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Number of Participants for Dose 200 mg: All participants received Acyclovir Tablet 200 mg with 240 mL of water (new and marketed)
- Total Number of Participants for Dose 400 mg: All participants received Acyclovir Tablet 400 mg with 240 mL of water (new and marketed)
- Total: Total of all reporting groups
Arm/Group | Total Number of Participants for Dose 200 mg | Total Number of Participants for Dose 400 mg | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 18 | 21 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Parameter
Description: Maximum plasma concentration (Cmax)
Time Frame: before dosing (0 h) and at 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after dosing
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Acyclovir 200 mg Tablet: Participants received Acyclovir Tablet 200 mg with 240 mL of water
- Zovirax® 200 mg Tablet: Participants received Zovirax® Tablet 200 mg with 240 mL of water
- Acyclovir 400 mg Tablet: Participants received Acyclovir Tablet 400 mg with 240 mL of water
- Zovirax® 400 mg Tablet: Participants received Zovirax® Tablet 2x200 mg with 240 mL of water
Arm/Group | Acyclovir 200 mg Tablet | Zovirax® 200 mg Tablet | Acyclovir 400 mg Tablet | Zovirax® 400 mg Tablet
Number analyzed (Participants) | 26 | 26 | 28 | 28
ng/mL | 613.21 (244.06) | 675.58 (258.18) | 807.13 (278.85) | 882.89 (351.97)

2. Primary Outcome: Pharmacokinetics Parameter
Description: Area Under Curve from 0 to 24 hours (AUCt)
Time Frame: Predose at (0 h) and at 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours post dose
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Acyclovir 200 mg Tablet | Zovirax® 200 mg Tablet | Acyclovir 400 mg Tablet | Zovirax® 400 mg Tablet
Number analyzed (Participants) | 26 | 26 | 28 | 28
ng*h/mL | 3609.80 (1425.19) | 3865.20 (1339.05) | 4583.29 (1518.93) | 5088.28 (1758.74)

3. Secondary Outcome: Geometric Mean Ratio
Description: The ratio between maximum concentration of test drug and reference drug after drug administration
Time Frame: before dosing (0 h) and at 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after dosing
Measure: Geometric Mean (90% Confidence Interval); unit: percentage
Arm/Group | Acyclovir 200 mg Tablet | Zovirax® 200 mg Tablet | Acyclovir 400 mg Tablet | Zovirax® 400 mg Tablet
Number analyzed (Participants) | 26 | 26 | 28 | 28
percentage | 90.65 [82.69 to 99.37] | 90.65 [82.69 to 99.37] | 93.63 [84.85 to 103.33] | 93.63 [84.85 to 103.33]

4. Secondary Outcome: Geometric Mean Ratio
Description: The ratio between area under curve from 0 to 24 hours of test drug and reference drug
Time Frame: before dosing (0 h) and at 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after dosing
Measure: Geometric Mean (90% Confidence Interval); unit: percentage
Arm/Group | Acyclovir 200 mg Tablet | Zovirax® 200 mg Tablet | Acyclovir 400 mg Tablet | Zovirax® 400 mg Tablet
Number analyzed (Participants) | 26 | 26 | 28 | 28
percentage | 92.74 [86.04 to 99.96] | 92.74 [86.04 to 99.96] | 90.10 [80.80 to 100.48] | 90.10 [80.80 to 100.48]

ADVERSE EVENTS:
Time Frame: before dosing (0 h) at 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours after dosing
Description: [Not Specified]
Arm/Group | Acyclovir 200 mg Tablet | Zovirax® 200 mg Tablet | Acyclovir 400 mg Tablet | Zovirax® 400 mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/26 | 1/26 | 1/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir 200 mg Tablet (N=26) | Zovirax® 200 mg Tablet (N=26) | Acyclovir 400 mg Tablet (N=28) | Zovirax® 400 mg Tablet (N=28)
Headache, Dizzines (Nervous system disorders) | 1 (26) | 1 (26) | 1 (28) | 1 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT04988646/Prot_SAP_000.pdf